CLINICAL TRIAL: NCT04137237
Title: Hand & Wrist Pyrocarbon Implants Outcomes Clinical Study
Acronym: HaWPYC
Status: Recruiting | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: 1803-W-HAPYC-RM; 2019-A00536-51 (Other: ANSM)
Record Dates: First submitted 2019-10-18; First posted 2019-10-23 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Orthopedics
Keywords: Hand; Wrist; Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
HaWPYC is an international Post-Market Clinical Follow-up (PMCF) to collect post-market safety and performance data on commercially available Pyrocarbon (PyC) hand and wrist implants used in this study. Data may be used for Post-Market Surveillance, and regulatory requirements.

DETAILED DESCRIPTION:
The objective of this multicenter study is to collect preoperative, intraoperative, intermediate (approx. 2 years), mid-term (approx. 5 years), and long-term (approx. 10 years) postoperative data, on related clinical complications and clinical outcomes on the Sponsors market-approved hand and wrist Pyrocarbon implants, to demonstrate safety and performance of these implants in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time he/she receives the information and signs the informed consent (when applicable as per local regulatory requirements),
* Informed on the study and willing to sign an informed consent form approved by Institutional Review Board or Ethics Committee,
* Willing and able to comply with the requirements of the study protocol,
* For prospective inclusion: considered for treatment with one of PyC Hand/Wrist study implants (primary or revision surgery),
* For "ambispective" inclusion: must have undergone a Hand or Wrist arthroplasty with a PyC Hand/Wrist study implant before the date of first site initiation visit,

  * Follow-up visits (at least the last two) must be prospective,
  * Patient must have complete information available for each completed visit

Exclusion Criteria:

* Patient pertaining to one of the categories referred to as "vulnerable population" in the French Law (articles L. 1121-5 to L. 1121-8 of the French Public Health Code), or as "particularly vulnerable persons" in the Swiss Federal Law (Chapter 3, Sections 1 to 4 of CC 810.30 Federal Act on Research involving Human Beings - Human Research Act, HRA),
* Patient unable to comply with the study procedures based on the judgment of the investigator (e.g. cannot comprehend study questions, inability to keep scheduled assessment times),
* Any medical condition that could impact on the study outcomes functional signification at the investigator's discretion (e.g., neuropathy, allergy…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 417 patients will be enrolled (About 50 to 80 per implant type). Prospective patients: screening and surgery should occur after the First site initiation visit.
  "Ambispective" patients:
  * Screening and surgery occurred before the date of the first site initiation visit,
  * Follow-up visits (at least the last two) must be prospective (i.e: must occur after the date of the first site initiation visit),
  * Inclusions of consecutive patients,
  * Minimum available data must be available for each completed visit.
Sampling Method: Non-Probability Sample
Enrollment: 417 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Total QuickDASH average compared to the predefined Minimal Clinically Important Difference (MCID) | 24 months
  Demonstrate a superior (lower) total QuickDASH average by 24 months postoperatively compared to the predefined Minimal Clinically Important Difference (MCID) upper threshold of 36 points.
  QuickDash = Disabilities of the Arm, Shoulder and Hand), self-report questionnaire; 11 items to measure physical function and symptoms; items scored on a 1-5-point scale which is then transformed resulting in a score from 0 (least disability) to 100 (most disability).

SECONDARY OUTCOMES:
Change from baseline in Patient Satisfaction scores | up to 10 years
  Single, subjective question measuring patient satisfaction; assessed through 4 levels satisfaction: "Very Satisfied, Satisfied, Dissatisfied, and Very Dissatisfied".
Safety evaluation | up to 10 years
  Number of device associated and procedure associated adverse events
Implant Survivorship | up to 10 years
  Rates of revision surgeries; assessed using the Kaplan-Meyer analysis
Clinical assessment: change from baseline in QuickDash score | up to 10 years
  QuickDash = Disabilities of the Arm, Shoulder and Hand), self-report questionnaire; 11 items to measure physical function and symptoms; items scored on a 1-5-point scale which is then transformed resulting in a score from 0 (least disability) to 100 (most disability).
Clinical assessment: change from baseline in PRWE score | up to 10 years
  PRWE = Patient-rated Wrist Evaluation; patient reported outcome developed to assess pain in the wrist joint and functional difficulties in activities of daily living resulting from injuries affecting wrist joint area. 15-item questionnaire made of two subscales (pain and function), resulting in a score from 0 to 100; Less score = better outcome.
Clinical assessment: change from baseline in Strength score | up to 10 years
  Grip/grasp, tip and key pinch strength will be evaluated using a dynamometer.
Clinical assessment: change from baseline in Mobility score | up to 10 years
  Evaluation of mobility (movement amplitude and functionality) will be assessed through angle measurement, using a goniometer. Measured movements will be flexion/extension, radial deviation/ulnar deviation, pronation/supination, adduction/abduction, opposition.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma
Locations (4):
- France (3):
  - Clinique du Parc, Lyon
  - Espace Médical Vauban, Paris
  - Institut de la Main Nantes-Atlantique - Pôle Santé-Atlantique, Saint-Herblain
- Orthopedic Surgeon (Dr. med. Dietmar Bignion), Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No